CLINICAL TRIAL: NCT00377676
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Assess Safety and Tolerability During Treatment of Type 2 Diabetes (T2DM) With Usual Diabetes Therapy (UDT) and Either Cycloset or Placebo
Brief Title: Safety and Tolerability Study of Cycloset in Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VeroScience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 165-AD-04-03-US-1
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Bromocriptine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Diabetes Therapy plus placebo (Experimental): Usual diabetes therapy plus placebo
  Interventions: Drug: Usual Diabetes Therapy plus placebo
- Drug Cycloset (Experimental)
  Interventions: Drug: Cycloset

INTERVENTIONS:
Drug: Cycloset — Usual diabetes therapy plus Cycloset
  Other Names: bromocriptine mesylate
  Arms: Drug Cycloset
Drug: Usual Diabetes Therapy plus placebo — Placebo tablet taken orally once in the morning, beginning with one tablet daily, titrated up by 1 tablet each week to a maximum of 6 tablets daily
  Other Names: placebo
  Arms: Usual Diabetes Therapy plus placebo

SUMMARY:
Cycloset, a new quick-release oral formulation of bromocriptine mesylate, effectively reduces blood sugar by the proposed mechanism of reversing many of the metabolic alterations associated with insulin resistance and obesity by resetting central (hypothalamic) circadian organization of monoamine neuronal activities.

The primary analysis of this study will test the hypothesis that the rate of all-cause severe adverse events for those receiving usual drug therapy for diabetes management plus Cycloset is not greater than that for usual drug therapy plus placebo by more than an acceptable margin. While the primary purpose of this study is to establish the safety profile of Cycloset in type 2 diabetes, any potential positive cardiovascular benefits will be evaluated as well.

DETAILED DESCRIPTION:
Bromocriptine mesylate, an ergot derivative, is a sympatholytic dopamine D2 receptor agonist that can exert inhibitory effects on serotonin turnover in the central nervous system. It has been proposed that bromocriptine can reverse many of the metabolic alterations associated with insulin resistance and obesity by resetting central (hypothalamic) circadian organization of monoamine neuronal activities.

While Cycloset has demonstrated efficacy by reducing HbA1c, fasting and post-prandial glucose and fasting and post-prandial triglycerides, the relatively small numbers of individuals treated for type 2 diabetes during the controlled Phase III clinical trials of Cycloset did not allow for a full evaluation of the safety profile. Since persons with diabetes are already at higher risk for cardiovascular disease, it is important to examine more fully the spectrum of potential adverse or positive effects from Cycloset in a large sample of persons with diabetes. Accordingly, the present study is designed to investigate the clinical safety of treatment with Cycloset in a broad population of persons with type 2 diabetes.

To determine in subjects with type 2 diabetes mellitus receiving Usual Diabetes Therapy (UDT) consisting of either diet, oral hypoglycemic agents (OHA) (no more than 2), or insulin (with or without no more than 1 OHA) plus either Placebo or Cycloset:

1. Whether add-on therapy with Cycloset results in all-cause rate of serious adverse events, which are not higher than add-on therapy with Placebo.
2. Whether add-on therapy with Cycloset results in disease-specific rate of serious cardiovascular adverse events, which are not higher than add-on therapy with Placebo.

   While the primary purpose of this study is to establish the safety profile of Cycloset in type 2 diabetes, any potential positive cardiovascular benefits will be evaluated as well.

   Other clinical measures:
3. The impact (either positive or negative) of Cycloset on HbA1c, fasting plasma glucose, weight, triglycerides lipids, blood pressure and patient tolerability after 12 months of therapy.

Furthermore, Hba1c changes from baseline to 24 weeks between Cycloset and Placebo among subjects with a baseline Hba1c of >= 7.5% among the following subgroups:

A. Treated at baseline with any Oral hypoglycemic agent (OHA) including injectable insulin secretagogues B. Metformin plus or minus one OHA or injectable insulin secretagogue C. Sulphonylurea plus or minus one OHA or injectable insulin secretagogue D. Treated at baseline with Metformin and one sulphonylurea

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* age 30-80 years
* body mass index < 43 kg/m2
* HbA1c ≤ 10% for at least 12 weeks prior to screening
* stable diabetes therapeutic regimen consisting of either diet, oral hypoglycemic agents (no more than 2), or insulin (with or without no more than 1 oral hypoglycemic agent) for 4 weeks prior to randomization

Exclusion Criteria:

* Subject who had taken prescription sympathomimetic drugs within seven (7) days prior to the first screening visit. Prescription sympathomimetic drugs were not allowed for any period greater than ten (10) consecutive days during the course of the study. Other ergot alkaloid derivatives or anti-migraine medications such as zolmitriptan (Zomig) and sumatriptan (Imitrex) were not permitted during the study.
* Subject who had a history of alcoholism or drug abuse in the three (3) years prior to the first screening visit.
* Subject who had a known hypersensitivity to any of the formulation components of the study drug.
* Subject who had received any experimental drug or used an experimental device in the 30 days prior to the first screening visit or would do so during the study.
* Subject who was pregnant or lactating women or women planning to become pregnant during the study. Women of childbearing potential had to have a negative pregnancy test at screening. Women who became pregnant were discontinued from the study.
* Subject who had given donations of blood during the 30 days prior to the screening visit. Donation of blood also was prohibited during the study and for 30 days after completion of the study.
* Subjects with clinically significant major organ system disease, such as

  * seizure disorder
  * significant gastroparesis or orthostatic hypotension (autonomic neuropathy)
  * cerebrovascular accident in the previous 6 months
  * uncontrolled hypertension (systolic BP >160 or diastolic BP > 100 at screening)
  * coronary artery bypass graft or coronary angioplasty in the previous 3 months, myocardial infarction in the previous 6 months, or unstable angina pectoris (chest pain at rest, worsening chest pain, or admission to the ER or hospital for chest pain) within the previous 3 months
  * congestive heart failure defined by NYHA as Class III or IV
  * clinical nephrotic syndrome, or renal impairment with a serum creatinine > 1.4 mg/dl if female receiving treatment with metformin, > 1.5 mg/dl if male receiving treatment with metformin, and > 1.6 mg/dl in not on metformin
  * impaired liver function, including having AST or ALT greater than three times the upper limit of normal
  * active infection (e.g., HIV, hepatitis), or a history of severe infection during the 30 days prior to screening
  * major surgical operation during the 30 days prior to screening
  * cancer, other than non-melanoma skin or non metastatic prostate cancer within the past 5 years
  * Any concurrent illness, other than diabetes mellitus, not controlled by a stable therapeutic regimen
* Working rotating, varying or night shifts
* Patients taking unapproved herbal supplements that may be associated with a risk of cardiovascular events (such as ephedra, yohimbe etc)
* Patients who had started therapy with an erectile dysfunction drug within 2 weeks prior to screening; patients could not begin treatment with an erectile dysfunction drug during the study period; patients previously taking erectile dysfunction drugs could do so only under medical supervision.
* Subjects with circumstances or abnormalities (e.g., blindness or a history of non-compliance) that would interfere with the interpretation of safety or efficacy data or completion of the study.
* Clinically significant abnormalities (values outside the normal range) on screening central laboratory evaluation unless discussed with and approved by the study principal investigator or Sponsor medical monitor.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3095 (Actual)
Dates: Start 2004-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gaziano, Principal Investigator — MAVERIC; Richard E Scranton, MD MPH, Principal Investigator — VeroScience

REFERENCES:
- [Background] Scranton RE, Gaziano JM, Rutty D, Ezrokhi M, Cincotta A. A randomized, double-blind, placebo-controlled trial to assess safety and tolerability during treatment of type 2 diabetes with usual diabetes therapy and either Cycloset or placebo. BMC Endocr Disord. 2007 Jun 25;7:3. doi: 10.1186/1472-6823-7-3. PMID 17592632
- [Result] Gaziano JM, Cincotta AH, O'Connor CM, Ezrokhi M, Rutty D, Ma ZJ, Scranton RE. Randomized clinical trial of quick-release bromocriptine among patients with type 2 diabetes on overall safety and cardiovascular outcomes. Diabetes Care. 2010 Jul;33(7):1503-8. doi: 10.2337/dc09-2009. Epub 2010 Mar 23. PMID 20332352
- [Derived] Chamarthi B, Cincotta AH. Effect of bromocriptine-QR therapy on glycemic control in subjects with type 2 diabetes mellitus whose dysglycemia is inadequately controlled on insulin. Postgrad Med. 2017 May;129(4):446-455. doi: 10.1080/00325481.2017.1315290. Epub 2017 Apr 12. PMID 28374645
- [Derived] Chamarthi B, Ezrokhi M, Rutty D, Cincotta AH. Impact of bromocriptine-QR therapy on cardiovascular outcomes in type 2 diabetes mellitus subjects on metformin. Postgrad Med. 2016 Nov;128(8):761-769. doi: 10.1080/00325481.2016.1243003. Epub 2016 Oct 11. PMID 27687032
- [Derived] Chamarthi B, Gaziano JM, Blonde L, Vinik A, Scranton RE, Ezrokhi M, Rutty D, Cincotta AH. Timed Bromocriptine-QR Therapy Reduces Progression of Cardiovascular Disease and Dysglycemia in Subjects with Well-Controlled Type 2 Diabetes Mellitus. J Diabetes Res. 2015;2015:157698. doi: 10.1155/2015/157698. Epub 2015 Apr 28. PMID 26060823
- [Derived] Gaziano JM, Cincotta AH, Vinik A, Blonde L, Bohannon N, Scranton R. Effect of bromocriptine-QR (a quick-release formulation of bromocriptine mesylate) on major adverse cardiovascular events in type 2 diabetes subjects. J Am Heart Assoc. 2012 Oct;1(5):e002279. doi: 10.1161/JAHA.112.002279. Epub 2012 Oct 25. PMID 23316290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 74 centers across the United States and Puerto Rico, including 19 Veterans Affairs (VA) hospitals. First patient enrolled: 23 August 2004 Last patient completed: 25 January 2007
Pre-assignment Details: 4,074 subjects were screened, 3,095 randomized 2:1 to Cycloset or placebo. 3,095 were analyzed for safety and 3,070 for all other analyses.The most common reason given for screen failure due to protocol ineligibility was an elevated creatinine (24.7% of all screen failures).
Groups:
- Cycloset: During the first week of the dose titration period, subjects were instructed to take 1 tablet of study drug daily (0.8 mg Cycloset). If the dose was tolerated, subjects were to have their dose of study drug increased to 2 tablets of study drug per day. The daily dose of study drug was to be increased at a rate of 1 tablet per week, up to a target dose level of 6 tablets per day at Week 6.
- Placebo: During the first week of the dose titration period, subjects were instructed to take 1 tablet of study drug daily (1 placebo tablet). If the dose was tolerated, subjects were to have their dose of study drug increased to 2 tablets of study drug per day. The daily dose of study drug was to be increased at a rate of 1 tablet per week, up to a target dose level of 6 tablets per day at Week 6.
Period: Overall Study
Arm/Group | Cycloset | Placebo
Started | 2054 (25 subjects did not receive study drug - thus 3070 were randomized and received drug) | 1016
Completed | 1093 | 694
Not Completed | 961 | 322
Not completed — Adverse Event | 498 | 107
Not completed — Protocol Violation | 33 | 27
Not completed — Death | 5 | 2
Not completed — Withdrawal by Subject | 187 | 72
Not completed — Lost to Follow-up | 120 | 56
Not completed — Other | 118 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cycloset | Placebo | Total
Number analyzed (Participants) | 2054 | 1016 | 3070
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1453 | 701 | 2154
  >=65 years | 601 | 315 | 916
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (10) | 59.5 (10) | 59.7 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 913 | 418 | 1331
  Male | 1141 | 598 | 1739
Region of Enrollment [Number; unit: participants]
  United States | 2054 | 1016 | 3070

OUTCOME MEASURES:

1. Primary Outcome: Subjects Experiencing Serious Adverse Events
Description: Number of subjects reporting all-cause Serious Adverse Events (SAEs) for usual drug therapy plus Cycloset vs. that for usual drug therapy (UDT) plus placebo from baseline to week 52.
Time Frame: From baseline to week 52.
Measure: Number; unit: participants
Arm/Group | Cycloset | Placebo
Number analyzed (Participants) | 2054 | 1016
participants | 176 | 98
Statistical Analysis 1: Comparison: Cycloset vs Placebo; Test type: Non-Inferiority or Equivalence — In order to test the primary hypothesis at a one-sided alpha = .05 and have a power of 0.9, when the non-inferiority margin is 1.5, the total number of subjects with all-cause SAEs that must be observed during the study was found to be 235. Assuming the placebo rate is 0.08, the required sample size was found to be 2991; p < 0.05, Regression, Cox — Using the Lan and Demets alpha spending function for O'Brien-Fleming boundaries and the overall one-sided significance level of 5%, a level of 0.04068 was to be used at the interim analysis and 0.03938 at the time of the final analysis; Hazard Ratio (HR) = 1.02, 95% CI 1-sided [upper limit 1.27] — cycloset to placebo

2. Secondary Outcome: Number of Subjects Experiencing Serious Cardiovascular Adverse Events
Description: The secondary safety endpoint is number subjects with occurrences of first cardiovascular SAE (myocardial infarction, stroke, in-patient hospitalization for heart failure, angina or revascularization surgery).
Time Frame: Baseline to week 52.
Population: intent to treat
Measure: Number; unit: Subjects
Arm/Group | Cycloset | Placebo
Number analyzed (Participants) | 2054 | 1016
Subjects | 31 | 30
Statistical Analysis 1: Comparison: Cycloset vs Placebo; In order to test the hypothesis for serious cardiovascular adverse events as for the primary endpoint at a one-sided alpha = 0.5 when the non-inferiority margin is 1.5, the final sample size of 3000 to 3300 subjects was to provide at least 62% power, assuming a hypothetical rate of events of 3.43%, or 103 to 113 cardiovascular SAEs. Upon demonstration of non-inferiority - a 2 sided using 95% CI was used to assess for superiority; Test type: Superiority or Other; p < 0.05, Regression, Cox; Cox Proportional Hazard = .58, 95% CI 2-sided [.35 to .96]

3. Secondary Outcome: Change in HbA1c From Baseline to Week 24 in Subjects Failing Treatment With Metformin Plus a Sulfonylurea
Description: Change in HbA1c from baseline to week 24 in subjects failing treatment with metformin plus a sulfonylurea with failure defined as having a baseline HbA1c value of ≥ 7.5%. Change was measured at week 24 after randomization in subjects having no major protocol violations.
  Change is reported as the absolute difference in % HbA1c.
Time Frame: Baseline to week 24
Population: subjects with baseline HbA1c of >= 7.5 and taking both metformin/sulfonylurea but not insulin. Analysis was conducted for those completing 24 weeks of treatment and on the ITT using the LOCF for those not completing 24 weeks of treatment.
Measure: Least Squares Mean (Standard Deviation); unit: percent
Arm/Group | Cycloset | Placebo
Number analyzed (Participants) | 177 | 90
percent | -0.49 (0.8) | -0.04 (1)
Statistical Analysis 1: Comparison: Cycloset; If the standard deviation of HbA1c level is about 1.0% and the baseline and 24 week scores have a correlation of 0.50 then the effect size is 0.5%/1.0% = 0.50. For the metformin/SU analysis, 160 subjects assuming a standard deviation of 1.0% would provide a power of 90% power to detect differences in mean changes of 0.5% or larger; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.5, Standard Deviation 1.4

4. Secondary Outcome: Change in HbA1c From Baseline to Week 24 for Subjects With a Baseline HbA1c of ≥ 7.5% Who Were Taking at Least One Oral Hypoglycemia Agent (OHA) at Baseline.
Description: The difference between Cycloset and placebo in the change in HbA1c from baseline to Week 24 was analyzed for subjects with a baseline HbA1c of ≥ 7.5% who were taking at least one oral hypoglycemia agent (OHA) at baseline. The primary analysis was based on subjects from the evaluable per protocol efficacy (EPPE) analysis set with a secondary analysis using subjects from the intent to treat efficacy (ITTE) analysis set for subjects completing 24 weeks of treatment. Change is reported as the absolute difference in % HbA1c.
Time Frame: Baseline to week 24
Population: randomized subjects with a baseline HbA1c of >= 7.5 taking one or two oral diabetes agents (not insulin)
Measure: Least Squares Mean (Standard Deviation); unit: percent
Arm/Group | Cycloset | Placebo
Number analyzed (Participants) | 261 | 151
percent | -0.41 (0.9) | 0.041 (1.2)
Statistical Analysis 1: Comparison: Cycloset vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.5

ADVERSE EVENTS:
Time Frame: Expected study duration was 52 weeks. Adverse event data were collected from the day of first treatment dose to within 30 days of the last course of treatment or the date of the last contact (whichever was earlier).
Arm/Group | Cycloset | Placebo
Serious Adverse Events (participants affected / at risk) | 176/2054 | 98/1016
Other Adverse Events (participants affected / at risk) | 1611/2054 | 430/1016
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycloset (N=2054) | Placebo (N=1016)
Cardiac Disorders (Cardiac disorders) | 51 (51) | 37 (37) — Cardiac Disorders include: Coronary Artery Disease, Chest Pain, Cardiac failure congestive, Myocardial Infarction, Angina Unstable, Atrial Fibrillation, Syncope, Acute Myocardial Infarction
Infection (Infections and infestations) | 27 (27) | 13 (13) — Infection includes: Pneumonia, Cellulitis, Diverticulitis
Nervous (Nervous system disorders) | 26 (26) | 14 (14) — Nervous system disorders include: Syncope, Cerebrovascular accident, Transient ischemic attack
General disorders and adminstrative site conditions (General disorders) | 14 (14) | 9 (9) — General disorders and administrative site conditions include: Chest pain, non-cardiac chest pain
Gastrointestinal (Gastrointestinal disorders) | 13 (13) | 9 (9) — Gastrointestinal disorders include: Gastrointestinal hemorrhage
Vascular disorders (Vascular disorders) | 10 (10) | 8 (8) — Vascular disorders include: Carotid artery stenosis
Respiratory (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 3 (3) — Respiratory, thoracic and mediastinal disorders include: Chronic obstructive pulmonary disease
Injury (Injury, poisoning and procedural complications) | 12 (12) | 3 (3)
Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 11 (11) | 4 (4)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 2 (2)
Endocrine disorders (Endocrine disorders) | 5 (5) | 4 (4) — Endocrine disorders include: hypoglycemia
Metabolism (Metabolism and nutrition disorders) | 7 (7) | 2 (2) — Metabolism and nutrition disorders include: Dehydration
Renal (Renal and urinary disorders) | 6 (6) | 3 (3) — Renal and urinary disorders include: acute renal failure
Hepatobiliary (Hepatobiliary disorders) | 4 (4) | 1 (1)
Pyschiatric (Psychiatric disorders) | 4 (4) | 1 (1)
Reproductive (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Eye (Eye disorders) | 0 (0) | 2 (2) — Eye disorders include: retinal detachment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycloset (N=2054) | Placebo (N=1016)
nausea (Gastrointestinal disorders) | 661 (661) | 77 (77)
vomiting (Gastrointestinal disorders) | 167 (167) | 32 (32)
Dizziness (Nervous system disorders) | 303 (303) | 63 (63)
headache (Nervous system disorders) | 235 (235) | 84 (84)
Fatigue (General disorders) | 285 (285) | 68 (68)
constipation (Gastrointestinal disorders) | 119 (119) | 52 (52)
hypoglycemia (Endocrine disorders) | 141 (141) | 54 (54)

LIMITATIONS AND CAVEATS:
Thus HbA1c was only performed on a subset of patients defined as failing (HbA1c >= 7.5) and who were on oral diabetes medications. Forced titration of study drug may have lead to a greater number of discontinuations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After FDA filing, Principal Liaison shall be free to publish the results of the Study subject only to the provisions of Section 7 regarding Veroscience Proprietary Information. The Principal Liaison shall furnish Veroscience with a copy of any proposed publication for review and comment prior to submission for publication, at least thirty (30) days prior to submission for manuscripts and at least fifteen (15) days prior to submission for abstracts.